CLINICAL TRIAL: NCT01374828
Title: Prospective Randomized Double-blind Study of Incisional Local Anesthesia in Laparoscopic Surgery (Ketorolac Versus Normal Saline)
Brief Title: Ketolorac Versus Saline at Laparoscopic Incision Sites
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 11-452
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Pain, Postoperative
Keywords: Toradol; Ketorolac; Normal saline; Laparoscopic; Postoperative pain control; Incisional analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketolorac (Experimental)
  Interventions: Drug: Ketolorac

INTERVENTIONS:
Drug: Ketolorac — Ketorolac 30 mg in 10 ml saline will be injected at the incision sites at the conclusion of the procedure.
  Other Names: Toradol

SUMMARY:
Pain control following surgery is a critical aspect of patient care. Pain at incision sites in laparoscopic surgery contributes to overall pain felt by a patient. There is no definitive proof that the typical medications (such as lidocaine) injected at incision sites during surgery improve pain control. This study looks at a different type of medication (ketorolac - an NSAID) to better control pain at laparoscopic incision sites.

DETAILED DESCRIPTION:
As the push for more minimally invasive and economical procedures increases, special attention will be paid to reasons why patients experience complications, unanticipated outpatient visits or require prolonged recovery times or even unplanned hospital admissions. Insufficient pain control is one of the prime reasons for increased level of care (16, 17), with pain defined as a "conscious unpleasant sensory and emotional experience associated with actual or potential tissue damage" (12). Appropriate pain control may advantageously affect length of hospital stay and related expense, decrease chronic pain syndromes, improve patient experience and result in fewer complications in the postoperative period (12).

Multiple methods of analgesia are employed to improve pain control after procedures, including intravenous medications, regional anesthesia and local injections (12, 16, 17). Laparoscopic procedures typically involve general anesthesia, and in an effort to improve recovery in the post anesthesia care unit (PACU) anesthesiologists employ shorter acting agents (2). Patients who received short acting anesthetic agents were more likely to bypass the PACU, particularly patients undergoing gynecologic surgery (2). This does not alleviate, and in fact may intensify, the need for adequate pain control in the immediate postoperative period.

Several strategies have been tested in an effort to improve analgesia in this critical time period, including intravenous, regional and local anesthesia (12). Multiple types of pain medications have been used to improve postsurgical pain. Opioids are commonly used, however may be associated with multiple negative affects including nausea and vomiting, delayed gastric emptying, sedation and respiratory depression (12). Postoperative nausea and vomiting, pain control and drowsiness were all factors contributing to prolonged recovery room stays (15). Other medications may be used to decrease opioid consumption, even the most common analgesics. Acetaminophen has been found to decrease opioid requirements postoperatively up to 20% (12). Postoperative NSAID use is quite common (12). With respect to NSAIDs in particular, ketorolac has been utilized due to its ability to improve pain control and lessen the amount of opioid medication given (12). Ketorolac offers advantages over opioids, particularly with respect to avoidance of and decrease in opioid associated side effects (4). These advantages have implications for both patient comfort and length of hospital stay following surgery. The use of adjunct non-opioid medications may lead to shorter PACU stays, decreased discharge times and fewer adverse effects such as respiratory depression and postoperative nausea and vomiting (4, 5, 15). Cassinelli et al demonstrated improved pain control when using IV ketorolac following lumbar decompression surgery, showing patients had decreased morphine requirements with improved pain scores following surgery. Coloma et al compared intravenous versus local ketorolac versus normal saline following anorectal surgery and found use of ketorolac in any form decreased pain scores. This was clinically significant in that it decreased the requirement for oral pain medications without a concomitant increase in side effects or complications. That group found that although both IV and local ketorolac provided pain relief following surgery, only local administration gave statistically significant lower pain scores on arrival to the PACU and had a shorter time to discharge compared to controls. In addition, a study by Ben-David found administration of 30 mg ketorolac locally had improved pain scores than when 60 mg was given intramuscularly (22). A comparison during orthopedic surgery of local vs systemic administration of ketorolac showed improved pain scores with local administration (23). These beneficial findings were in no way universal. Kardash et al compared ketorolac use in patients undergoing hernia repair and found no difference in pain levels postoperatively whether patients had ketorolac injected either at the site of the incision or peripherally (in this case a subcutaneous injection in the contralateral abdominal wall). These findings were mitigated somewhat due to lack of a control group, omitted primarily because the authors felt NSAIDs were a routine part of postoperative pain control and could not be ethically withheld. Ketorolac does have drawbacks in the form of suspected hematologic impact affecting platelet aggregation and bleeding time and must be used with cautiously in patients with renal compromise (12).

The source of pain is multifactorial, including not only intra-abdominal discomfort from the procedure itself but also from the skin incision as well (3). Multiple studies have compared local anesthesia injected at the site of laparoscopic incision to a normal saline control. Khaira et al examined normal saline vs. bupivacaine injections at the surgical incision site early in surgery and found a decrease in parenteral opioid use in patients who received the anesthetic injection. Cansino et al compared oral NSAID combined with a lidocaine paracervical block to oral placebo and a paracervical block that included both lidocaine and ketorolac during first trimester surgical abortion. They found improved pain control with the combined paracervical block particularly during cervical dilation, although the remaining pain scores were not significantly different. Mohair et al examined the effects of infiltration with pain medication in postoperative pain control in patients undergoing breast augmentation. They did this by infiltrating normal saline, ketorolac, bupivacaine or both ketorolac and bupivacaine into the breast pocket following dissection. Their results suggested the combined medication improved pain levels immediately postoperative and through the time of discharge at their outpatient surgery center. Each pain medication alone also improved pain scores although to a lesser extent. It is unclear if the statistical significance translates to a clinical significance. A follow up to the initial study of pain medication infiltrated into breast pockets in breast augmentation followed longer term pain scores in postoperative patients who had either normal saline or the combination ketorolac and bupivacaine infiltrated during surgery. Results showed improved pain scores over the first five postoperative days as determined by the visual analogue scale and amount of pain medication used when the analgesic solution was infiltrated during surgery. Again, it remains unclear whether this is clinically significant, as the amount of pain medication utilized differed by approximately one to two tablets daily. Mahabir et al theorized the possible benefit of ketorolac over bupivacaine could stem from the difference in pKa in the two medications. The pKa of ketorolac is 3.5, indicating a higher activity in acidic tissues, such as those that are damaged and inflamed, relative to a medication such as bupivacaine with its more basic pKa of 8.1 (16).

Not only is the type of analgesia in question but also the timing in administration: preincisional vs. at surgical closure. Einarsson et al specifically investigated local pain control in laparoscopic port sites using patients as their own controls. This study compared pain control in patients with bupivacaine and normal saline infiltrated at port sites, using each patient as their own control and found postoperative administration of bupivicaine resulted in better pain control. Ke et al examined efficacy of pain control with respect to both medication administered as well as timing when they compared infiltration of wounds with either bupivacaine or normal saline before initial incision or at incision closure. The results indicated pre-incision injection provided better pain control with longer lasting analgesic effects, however the study was limited by a small sample size leading to possibly less significant results. Lam et al also investigated local pain control at laparoscopic port sites with a placebo controlled trial using either lignocaine or normal saline at the initial incision or at closing the case. Their results advocated for using analgesia at the time of closure, showing decreased pain scores for up to 24 hours postoperatively in that group, and only minimal improvement with preemptive analgesia. These results may not be clinically significant because despite the decreased pain scores, amount of pain medication utilized was the same. Despite some studies indicating improved pain control with local anesthesia, multiple randomized, placebo controlled, double blind studies have not shown any significant difference between saline and bupivacaine with respect to post operative pain (18-21).

ELIGIBILITY:
Inclusion Criteria:

* Female undergoing gynecologic laparoscopic surgery
* Surgeries less than 60 minutes

Exclusion Criteria:

* Patients with a diagnosis of stage III or IV endometriosis, chronic pelvic pain, chronic narcotic use, allergy to anesthetics, contraindication to ketolorac
* Robotic assisted procedures, single-port laparoscopy or conversion to laparotomy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determine if ketorolac decreases incisional pain in laparoscopic surgery | 60 minutes post-op, 120 minutes post-op, at D/C from PACU and 24-hours following surgery

SECONDARY OUTCOMES:
Determine if amount of postoperative narcotics decreases after ketorolac use; monitor side effects and adverse outcomes | 60-minutes post-op; 120 minutes post-op; at time of D/C from PACU; and 24-hours post-op

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Goldberg, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic - Beachwood Ambulatory Surgery Center, Beachwood, Ohio, United States